CLINICAL TRIAL: NCT05970289
Title: A Phase 2 Multicenter, Randomized, Open-label Study to Investigate the Efficacy and Safety of BRII-835 (VIR-2218) and Pegylated Interferon Alpha (PEG-IFNα) Combination Therapy for the Treatment of Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Investigate the Efficacy and Safety of BRII-835 (VIR-2218) and PEG-IFNα Combination Therapy in Chronic HBV Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRII-835-002
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (Experimental): Participants will receive multiple doses of PEG-IFNα for 48 weeks.
  Interventions: Biological: PEG-IFNα
- Cohort 2 (Experimental): Participants will receive multiple doses of higher dose level of BRII-835 + PEG-IFNα for 48 weeks.
  Interventions: Biological: PEG-IFNα; Drug: BRII-835
- Cohort 3 (Experimental): Participants will receive multiple doses of lower dose level of BRII-835 + PEG-IFNα for 48 weeks.
  Interventions: Biological: PEG-IFNα; Drug: BRII-835
- Cohort 4 (Experimental): Participants will receive multiple doses of lower dose level of BRII-835 + PEG-IFNα for 48 weeks (participants who received BRII-179 in a previous study will roll over into this cohort).
  Interventions: Biological: PEG-IFNα; Drug: BRII-835

INTERVENTIONS:
Biological: PEG-IFNα — PEG-IFNα will be given via subcutaneous injection
  Other Names: pegylated interferon alfa
Drug: BRII-835 — BRII-835 will be given via subcutaneous injection
  Arms: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
This study will evaluate the efficacy and safety of PEG-IFNα alone or in combination with different dose levels of BRII-835 (VIR-2218) in participants with chronic hepatitis B virus (HBV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60.
* Body mass index ≥ 18 kg/m2 and ≤ 32 kg/m2.
* Chronic HBV infection for ≥ 6 months.
* On NRTI therapy for at least 6 months.

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the participant unsuitable for participation.
* Significant liver fibrosis or cirrhosis.
* History or evidence of drug or alcohol abuse.
* History of intolerance to SC injection.
* History of chronic liver disease from any cause other than chronic HBV infection.
* History of hepatic decompensation.
* Contraindications to the use of Peg-IFNα.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HBsAg loss at end of treatment | Up to Week 48
Proportion of participants with HBsAg loss at 24 weeks post-end of treatment | Up to Week 72
Proportion of participants with treatment-emergent adverse events (TEAEs) | Up to Week 72
Proportion of participants with serious adverse events (SAEs) | Up to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Chen, Study Director — Brii Biosciences Limited
Locations (28):
- Australia (3):
  - Investigative Site 61001, Kingswood, New South Wales
  - Investigative Site 61002, Birtinya, Queensland
  - Investigative Site 61003, Melbourne, Victoria
- China (12):
  - Investigative Site 86001, Beijing, Beijing Municipality
  - Investigative Site 86007, Beijing, Beijing Municipality
  - Investigative Site 86004, Chongqing, Chongqing Municipality
  - Investigative Site 86006, Guangzhou, Guangdong
  - Investigative Site 85201, Hong Kong, HONG KONG
  - Investigative Site 85202, Hong Kong, HONG KONG
  - Investigative Site 86008, Changchun, Jilin
  - Investigative Site 86013, Shanghai, Shanghai Municipality
  - Investigative Site 88601, Kaohsiung, Taiwan
  - Investigative Site 88602, Taipei, Taiwan
  - Investigative Site 88603, Taipei, Taiwan
  - Investigative Site 86011, Hangzhou, Zhengjiang
- Singapore (2):
  - Investigative Site 65001, Singapore
  - Investigative Site 65002, Singapore
- South Korea (6):
  - Investigative Site 82002, Chuncheon, Chuncheon-si
  - Investigative Site 82001, Busan
  - Investigative Site 82004, Daegu
  - Investigative Site 82005, Seoul
  - Investigative Site 82003, Seoul
  - Investigative Site 82006, Soeul
- Thailand (5):
  - Investigative Site 66003, Bangkok
  - nvestigative Site 66007, Chiang Mai
  - Investigative Site 66005, Khon Kaen
  - Investigative Site 66006, Nonthaburi
  - Investigative Site 66008, Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong GL, Yuen MF, Lin B, Douglas MW, Hu P, Xie Q, Lv F, Tak WY, Leerapun A, Kim DJ, Tangkijvanich P, Lim YS, Dai CY, O'Beirne J, Weltman M, Khemnark S, Piratvisuth T, Manasirisuk W, Chen X, Liu CJ, Heo J, Lee J, Niu J, Kumar R, Kumar R, Zhu C, Cao K, Tian A, Chen X, Zhu Q, Margolis D, Jia J, Hong Z. Elebsiran and PEG-IFNalpha for chronic hepatitis B infection: a partially randomized, open-label, phase 2 trial. Nat Med. 2026 Jan;32(1):151-159. doi: 10.1038/s41591-025-04049-z. Epub 2025 Nov 7. PMID 41203919